CLINICAL TRIAL: NCT03027674
Title: "Color Doppler Ultrasound Comparison of Topical 10 % Nifedipine Versus 5% Sildenafil in Secondary Raynaud: A Randomized, Double-blind, Placebo-controlled Pilot Study"
Brief Title: Topical 10 % Nifedipine Versus 5% Sildenafil in Secondary Raynaud
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-234
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Raynaud Phenomenon Due to Trauma; Raynaud Disease; System; Sclerosis; Lupus Erythematosus, Systemic; Dermatomyositis; Ultrasound Therapy; Complications
Keywords: Raynaud Phenomena; System; Sclerosis; Lupus Erythematosus, Systemic; Ultrasound; sildenafil; Nifedipine
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse; Lupus Erythematosus, Systemic; Dermatomyositis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10% nifedipine cream (Experimental): Patient hands (right versus left) were randomized to treatment with topical sildenafil or nifedipine cream. The thumbs of both hands didn't receive any cream so that each subject served as her own control. Subjects were instructed to apply 5 grams of 10% nifedipine cream in one hand and 5 grams of 5% sildenafil cream to the opposite hand. Vinyl gloves were supplied to improve the absorption of the cream into the hand, leaving the thumb of both hands out of the glove without any cream.
  Interventions: Drug: 10% nifedipine cream
- 5% sildenafil cream (Active Comparator): Patient hands (right versus left) were randomized to treatment with topical sildenafil or nifedipine cream. The thumbs of both hands didn't receive any cream so that each subject served as her own control. Subjects were instructed to apply 5 grams of topical10% nifedipine cream in one hand and 5 grams of topical 5% sildenafil cream to the opposite hand. Vinyl gloves were supplied to improve the absorption of the cream into the hand, leaving the thumb of both hands out of the glove without any cream.
  Interventions: Drug: 5% sildenafil cream

INTERVENTIONS:
Drug: 10% nifedipine cream — Topical treatment for Raynaud
  Other Names: Topical treatment for Raynaud
  Arms: 10% nifedipine cream
Drug: 5% sildenafil cream — Topical treatment for Raynaud
  Other Names: Topical treatment for Raynaud
  Arms: 5% sildenafil cream

SUMMARY:
Objective: To compare the efficacy of topical 10% nifedipine versus 5% sildenafil in patients with secondary Raynaud's phenomenon (RP).

Methods: A randomized, double-blind, placebo-controlled pilot study took place in 10 patients with secondary RP. Topical 10% nifedipine on one hand and 5% sildenafil on the other hand were applied. The thumbs didn't receive any cream and served as a control group. The primary outcome was the improvement of blood flow and vessel diameter of the digital arteries measured by high frequency color Doppler ultrasound before and 1 hour after treatment.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is an exaggerated vascular response characterized by at least biphasic change (pallor and cyanosis) in the skin color of the digits, induced by cold temperature or emotional stress, The prevalence varies from 3 to 5%. In primary RP, there is no evidence of a secondary cause and patients have a younger age at onset (between 15 and 30 years), whereas in secondary RP, patients are older and have a connective tissue diseases (CTD), such as systemic sclerosis (SSc), systemic lupus erythematosus (SLE), dermatomyositis (DM), Sjögren's syndrome and rheumatoid arthritis. In secondary RP there are endothelial dysfunction and intimal fibrosis that compromise capillary blood flow. The treatment includes maintaining warmth of the whole body, smoking cessation and avoiding cold exposure, sympathomimetic medications and emotional stress. When these measures fail, the first line drugs are calcium-channel blockers (CCBs), eg. nifedipine. If CCBs are ineffective or not tolerated, a phosphodiesterase type 5 inhibitor (PDE-5), eg. sildenafil, or a topical nitrate should be used alone or in combination with CCBs. Other drugs includes serotonin reuptake inhibitors, angiotensin receptor blockers and prostaglandins. Unfortunately, secondary RP in patients with CTD most often is refractory to standard therapies, becoming a therapeutic challenge for clinicians. Based on the pathophysiology, topical vasodilators may act as an adjuvant therapy. Several randomized trials have demonstrated the benefit of various forms of topical nitrates (eg. nitroglycerin). In relation to other topical agents, solid evidence is lacking. Color Doppler ultrasound is a noninvasive imaging method that allows observation with good definition of skin and deep planes, including vascularization in real time.

The aim of this study is to compare the efficacy of topical 10% nifedipine versus 5% sildenafil in patients with secondary RP using high-frequency color Doppler ultrasound Patients The inclusion criteria considered patients with secondary RP associated with a CTD diagnosed and under follow-up in the Department of Dermatology. Diagnosis of CTD was made according to the ACR classification criteria for SSc, the Mixed Connective Tissue Disease criteria proposed by Kasukawa et al, the Bohan and Peter DM criteria and the SLICC SLE criteria. The exclusion criteria were primary RP patients; concurrent infection of any digit; allergic reaction and current use of any CCB or PDE-5 inhibitor;, , pregnancy, hypo and hypertension, history of myocardial infarction, stroke, or life-threatening arrhythmia. All patients signed a written informed consent. The Ethics Committee of Pontificia Universidad Católica de Chile approved the study protocol.

Study design This prospective study was conducted in August 2016 (winter). After screening, patients who were being treated with a vasodilator were required to discontinue it for at least 24 hours before randomization. All patients were receiving immunosuppressive treatment for their underlying disease. Patient hands (right versus left) were randomized to treatment with topical sildenafil or nifedipine cream. The thumbs of both hands didn't receive any cream so that each subject served as her own control. Subjects were instructed to apply 5 grams of 10% nifedipine cream in one hand and 5 grams of 5% sildenafil cream to the opposite hand. Vinyl gloves were supplied to improve the absorption of the cream into the hand, leaving the thumb of both hands out of the glove without any cream.

Clinical assessments The temperature of the examination room was set at 19ºC (66ºF) for ≥ 30 min and all patients underwent a high-frequency color Doppler ultrasound examination before and 1 hour after the topical treatments. The same radiologist with extensive experience in dermatologic ultrasound, performed all sonographic examinations. The radiologist was blinded to the clinical data of the study and the senior dermatologist in charge of the supervision of the application of the topical treatments was blinded to the color Doppler ultrasound results. The ultrasound equipment was a Logic E9 XD Clear working with a high frequency (upper range 18 MHz) compact linear probe (General Electric Health Systems, Waukesha, WI). The ultrasound protocol included grey scale, color Doppler and spectral curve analysis of the arterial flow using the settings of the machine for studying skin and superficial structures. The ultrasound device automatically provided the values. The primary outcome was the improvement of blood flow in the digital arteries. For Doppler sonography, peak systolic velocity (PSV, cm/sec) and diameter (mm) were measured at the palmar proper digital (PPD) arteries (proximal phalanx level) of radial aspect of the index, middle and thumb fingers of both hands. Also, PSV and diameter were measured at the dorsal (PD) arterial arch of the proximal nail fold of the index, middle and thumb fingers of both hands. Immediate and late adverse effects were monitored in all patients until 3 months after the study.

Statistical analysis PSV of the PPD artery and PD arterial arch of the index and middle fingers were added for a total PSV. The diameter of the PPD artery and PD arterial arch of the index and middle fingers were added for a total diameter. Due to the low velocity ranges, the values of peak systolic velocities in cm/sec were transformed into mm/sec. Treatment efficacy was assessed by using the differences in digital artery blood flows (total PSV) and diameters (total diameter) at baseline (time [t] = 0) and after 60 minutes (t = 60). Difference in digital artery blood flow and the digital artery diameter was defined as (t = 0) minus (t = 60); thus, the efficacy of the treatment was reflected by a negative difference. In all cases, mean differences less than zero indicates that the study drug cream was effective; mean differences greater than or equal to zero indicates that the study drug cream was ineffective. The Wilcoxon signed-rank tests and paired t-tests were used to assess the changes in outcomes within the group before and after treatment as appropriate. All tests were performed using two-tailed probabilities and p ≤ 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of secondary Raynaud´s phenomenon associated with a connective tissue disease

Exclusion Criteria:

* Primary Raynaud´s phenomenon
* Current infection of any digit
* Known allergic reaction to calcium-channel blockers or phosphodiesterase type 5 inhibitor
* Current use of calcium-channel blockers or phosphodiesterase type 5 inhibitors
* Pregnancy
* Hypotension or hypertension
* History of myocardial infarction, stroke, or life-threatening arrhythmia.

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Improvement of blood flow in the digital arteries (peak systolic velocity ) of the dorsal arterial arch of the proximal nail fold of the index, middle and thumb fingers of both hands | Outcome measure will be assessed the same day of the study and the data will be presented after the data is analyzed (12 weeks)
  The peak systolic velocity peak is measured with Doppler sonography in centimeters/second

SECONDARY OUTCOMES:
Improvement of the diameter (mm) of the dorsal arterial arch of the proximal nail fold of the of the index, middle and thumb fingers of both hands. | Outcome measure will be assessed the same day of the study and the data will be presented after the data is analyzed (12 weeks)
  The diameter is measured with Doppler sonography in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Vera-Kellet, MD, Principal Investigator — Connective Tissue Diseases Unit, Department of Dermatology Facultad de Medicina, Pontificia Universidad Católica de Chile, Santiago, Chile.
Locations (1):
- Department of Dermatology, Facultad de Medicina, Pontificia Universidad Católica de Chile, Santiago, Chile., Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No